CLINICAL TRIAL: NCT00285428
Title: A Phase I Study of Immunotherapy With hA20 Administered Once Weekly for 4 Consecutive Weeks in Patients With CD20+ Non-Hodgkin's Lymphoma
Brief Title: Study of hA20 (Humanized Anti-CD20) in Patients With CD20+ Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: William Wegener, MD, PhD, Immunomedics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hA20-01; NCT00112970 (obsolete NCT alias)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2012-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: treatment; NHL; CD20+ B-cell NHL; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — veltuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose level 1 (Experimental): 120 mg/m2
  Interventions: Drug: hA20-humanized anti-CD20 antibody
- Dose level 2 (Experimental): 200 mg/m2
  Interventions: Drug: hA20-humanized anti-CD20 antibody
- Dose Level 3 (Experimental): 375 mg/m2
  Interventions: Drug: hA20-humanized anti-CD20 antibody
- Dose level 1B (Experimental): 80 mg/m2
  Interventions: Drug: hA20-humanized anti-CD20 antibody

INTERVENTIONS:
Drug: hA20-humanized anti-CD20 antibody — once weekly iv dosing for 4 weeks
  Other Names: veltuzumab; IMMU-106; hA20

SUMMARY:
This is a Phase I trial to look at safety and how a patient's body will tolerate the treatment at different dosages.

ELIGIBILITY:
Inclusion Criteria:

* CD20+ B-cell non-Hodgkin's lymphoma (NHL) with measurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance of different dose levels | 12 weeks

SECONDARY OUTCOMES:
Lack of immunogenicity | 8 and 12 weeks
Pharmacodynamics | over 12 weeks
Pharmacokinetics | over 12 weeks
Efficacy | 4, 8 and 12 wks, every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (3):
- United States (3):
  - New York Presbyterian Hospital/Cornell Medical Center, New York, New York
  - University Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Goldenberg DM, Morschhauser F, Wegener WA. Veltuzumab (humanized anti-CD20 monoclonal antibody): characterization, current clinical results, and future prospects. Leuk Lymphoma. 2010 May;51(5):747-55. doi: 10.3109/10428191003672123. PMID 20214444
- [Result] Morschhauser F, Leonard JP, Fayad L, Coiffier B, Petillon MO, Coleman M, Schuster SJ, Dyer MJ, Horne H, Teoh N, Wegener WA, Goldenberg DM. Humanized anti-CD20 antibody, veltuzumab, in refractory/recurrent non-Hodgkin's lymphoma: phase I/II results. J Clin Oncol. 2009 Jul 10;27(20):3346-53. doi: 10.1200/JCO.2008.19.9117. Epub 2009 May 18. PMID 19451441